CLINICAL TRIAL: NCT07376850
Title: Time in rANge vs. Time in nOrmal Glycemia for Better Glycemic Control
Acronym: TANGO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Motol (Other)
Collaborators: Schneider Children's Medical Center, Israel (Other); Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Zdeněk Šumník, MD, PhD, University Hospital, Motol
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TANGO
Record Dates: First submitted 2025-12-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Diabetes; Diabetes (DM); Diabetes Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insemination, Artificial, Heterologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIR group (Active Comparator): Participants in this group will follow the current standard international clinical guidelines, targeting a glycemic range of 3.9-10.0 mmol/L (70-180 mg/dL). They will receive the same level of structured multidisciplinary education and clinical follow-up as the intervention group, but calibrated to the standard 70-180 mg/dL range.
  Interventions: Other: Structured Diabetes Education
- TING group (Experimental): Participants in this group will target a tighter glycemic range of 3.9-7.8 mmol/L (70-140 mg/dL). Their CGM and insulin pump settings will be adjusted by their physician to support this narrower range. Participants will receive structured education focused on achieving this tighter target.
  Interventions: Other: Structured Diabetes Education; Other: Automated Insulin Delivery (AID) System Adjustment

INTERVENTIONS:
Other: Structured Diabetes Education — A comprehensive standardized guideline will be provided to recruiting physicians from all centers, including the points below:
  1. Understanding CGM data and trend interpretation
  2. TIR or TING concepts according to randomization, target range, consequences of hypoglycemia and hyperglycemia
  3. Recognizing and management of hypoglycemia
  4. Recognizing and management of hyperglycemia
  5. Setting and adjusting of glycemic targets, alarms in CGM and insulin pumps, and insulin doses based on randomisation
  6. Emotional coping strategies and involving family support
Other: Automated Insulin Delivery (AID) System Adjustment — For the TING group, CGM hyperglycemia target settings will be lowered by at-least 10% from the baseline values. The extent of the adjustment will be at the discretion of the attending physician
  Arms: TING group

SUMMARY:
The TANGO study is a 12-month study involving 120 children and adolescents with Type 1 Diabetes (T1D) across the Czech Republic, Israel, and Poland who use automated insulin delivery (AID) systems.

Currently, the global standard for diabetes management is "Time in Range" (TIR), which aims to keep blood sugar levels between 70-180 mg/dL. However, newer technologies like AID systems may now allow for a tighter, more physiological goal called "Time in Normal Glycemia" (TING), which targets a range of 70-140 mg/dL.

This study will randomly assign participants to follow either the standard TIR target or the tighter TING target to see if the narrower range improves overall blood sugar control and HbA1c without increasing the risk of hypoglycemia, family stress, or daily treatment burden.

By comparing these two approaches, researchers hope to determine if clinical guidelines should be updated to reflect a more precise glucose target for children and adolescents worldwide

DETAILED DESCRIPTION:
This multinational, multicenter, randomized controlled trial aims to evaluate the clinical impact of targeting Time in Normal Glycemia (TING; 70-140 mg/dL) compared to the current standard, Time in Range (TIR; 70-180 mg/dL), in children and adolescents with Type 1 Diabetes (T1D).

Background and Rationale Managing glucose levels in pediatric T1D is essential for preventing long-term complications. While the international consensus currently recommends maintaining a TIR >70%, recent technological advances-such as automated insulin delivery (AID) systems and next-generation continuous glucose monitors (CGM)-now make it feasible to target narrower, more physiological glucose ranges. TING (70-140 mg/dL) has emerged as a potential new clinical metric for improved metabolic compensation. However, there is no definitive evidence yet that aiming for this tighter range leads to better long-term outcomes than the standard TIR without increasing treatment burden or psychological stress.

Study Objectives The primary objective is to determine if setting TING as the glycemic target improves CGM-derived glycemic metrics compared to the standard TIR approach.

Secondary objectives include:

Evaluating changes in HbA1c. Assessing differences in Quality of Life (QoL) and treatment burden using standardized patient and caregiver questionnaires.

Monitoring the safety and incidence of acute complications, such as severe hypoglycemia and diabetic ketoacidosis (DKA).

Study Design and Population The study will enroll 120 children and adolescents (ages 5.0-17.99) across three tertiary pediatric diabetes centers in the Czech Republic, Israel, and Poland. All participants must be using AID systems and have used a CGM for at least 70% of the time in the month prior to enrollment.

From the target population, we aim to recruit 25% of individuals newly diagnosed.

Intervention and Methods

Participants will be randomized 1:1 into two groups:

TING Group (Intervention): Will follow a target glucose range of 70-140 mg/dL (3.9-7.8 mmol/L).

TIR Group (Control): Will follow the standard target range of 70-180 mg/dL (3.9-10.0 mmol/L).

Both groups will receive structured education from a multidisciplinary team regarding CGM interpretation, glycemic targets, and self-management. In the TING group, CGM hyperglycemia targets will be lowered by at least 10% from baseline.

Timeline and Endpoints The study duration is 12 months. Data collection includes CGM metrics, insulin dose data, and HbA1c at 3-month intervals (Months 0, 3, 6, 9, and 12). A telephone check-up will occur 6 weeks after baseline to assess early adherence and treatment satisfaction.

Primary Endpoint: Change in TIR (70-180 mg/dL) between baseline and 12 months.

Secondary/Exploratory Endpoints: Percentage of time in TING, time in hypoglycemia (Levels 1 and 2), glycemic variability, and various QoL scores (PAID, INSPIRE, Hypoglycemia/Hyperglycemia Fear Surveys) .

Impact If targeting TING is proven beneficial and acceptable, the results of this trial could inform future clinical guidelines and redefine optimal glycemic targets for pediatric diabetes care globally.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T1D per ADA criteria
* Age 5.0-17.99 at the start of study
* CGM use >70% of the time during the month prior to enrollment
* Maximum HbA1c of 86mmol/mol (10% in DCCT)

Exclusion Criteria:

* No concurrent illnesses impacting glycemia
* No treatments impacting glycemia
* Severe hypoglycemia documented in the 60 day period leading up to patient recruitment
* Current participation in any other interventional study
* Any significant diseases / conditions including psychiatric disorders and substance abuse that in the opinion of the investigator is likely to affect the subject's ability to complete the study or compromise participant's safety
* Female subject who is pregnant or lactating or planning to become pregnant within the planned study duration

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 12 months
  Change in TIR over 12 months (between M0 and M12) between TING and TIR groups

SECONDARY OUTCOMES:
Diabetes-Related Emotional Distress in Pediatric Participants (PAID-Teen | At enrollment, 6 months and 12 months
  A 20-item survey assessing emotional distress. Items are scored 0-4. Unit of Measure: Standardized score (Range: 0 to 100). Interpretation: Higher scores indicate higher distress.
Participant Perceptions of Diabetes Technology - INSPIRE Patient Scale | At enrollment, 6 months and 12 months
  QoL questionnaire: Assesses how young patients feel about their insulin delivery systems.
  Unit of Measure: Score on a scale (Range: 0 to 100). Higher scores indicate higher satisfaction and more positive expectations of the device.
Quality of Life (QoL) Related to Diabetes Technology - INSPIRE Parent/Caregiver Scale | At enrollment, 6 months and 12 months
  Assesses parent/caregiver perceptions of automated insulin delivery systems. Each item is scored 0-4.
  Unit of Measure: Score on a scale (Range: 0 to 100). Interpretation: Higher scores indicate a more positive appraisal of the technology and better QoL.
Parent/Caregiver Fear of Hypoglycemia (HFS-P) | At enrollment, 6 months and 12 months
  A 26-item survey with two subscales: Behavior (11 items) and Worry (15 items). Items are rated from 0 (never) to 4 (very often).
  Unit of Measure: Total score (Range: 0 to 104). Interpretation: Higher scores indicate a greater fear of hypoglycemia.
Parent/Caregiver Fear and Behaviors Related to Hyperglycemia (HAQ) | At enrollment, 6 months and 12 months
  QoL questionnaire: Measures the extent of potentially problematic attitudes and behaviors used to avoid high blood sugar. It consists of 22 items rated 0-4.
  Unit of Measure: Total score (Range: 0 to 88). Interpretation: Higher scores indicate greater levels of hyperglycemia-related worry and more frequent avoidance behaviors.
Diabetes-Related Emotional Distress in Parents/Caregivers (PAID-PR) | At enrollment, 6 months and 12 months
  A 18-item scale measuring the emotional burden of caregiving. Items are rated from 0 (no problem) to 4 (serious problem).
  Unit of Measure: Total score (Range: 0 to 72). Interpretation: Higher scores reflect greater diabetes-specific emotional distress.

OTHER OUTCOMES:
Exploratory endpoints | 12 months
  Difference in the percentage of time in range (TIR) and time in normal glycemia (TING) at 3, 6, 9, and 12 months
Exploratory endpoints | 12 months
  Change in time in hypoglycemia level 1 (3,0-3,8 mmol/l) and level 2 (<3,0 mmol/l), hyperglycemia level 1 (10,1-13,9 mmol/l) and level 2 (>13,9 mmol/l) at 3, 6, 9, and 12 months
Exploratory endpoints | 12 months
  Change in Glycemic variability (SD, CV)
Exploratory endpoint | 12 months
  Change in Mean glucose level
Exploratory endpoint | 12 months
  Difference in Insulin dose
Exploratory endpoint | 12 months
  Change in HbA1c

CONTACTS AND LOCATIONS:
Locations (3):
- Motol University Hospital, Prague, Czechia
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel
- Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the anonymised participants' data on individual request
Supporting Information: Study Protocol